CLINICAL TRIAL: NCT05201898
Title: Dietary Intervention for Cardiovascular Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the severe epidemic situation of COVID-19 and the shortage of research funds and manpower for research projects, the study was halted prematurely.
Sponsor: Academia Sinica, Taiwan (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, Wen-Harn Pan, Distinguished Research Fellow, Principal Investigator, Academia Sinica, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AS-IRB-BM-19057
Record Dates: First submitted 2021-12-19; First posted 2022-01-21 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- usual medical management (Placebo Comparator): with regular doctor visits every 3 months
  Interventions: Other: control:usual medical management
- usual medical management+individual dietary consultation (Experimental): with regular doctor visits every 3 months and dietitian visits every 3 months until meeting dietary recommendation or reaching 3 years limit
  Interventions: Other: control:usual medical management; Behavioral: intervention 1:usual medical management+individual dieting consultation
- usual medical management+individual dietary consultation+ daily tea drinking (Experimental): with regular doctor visits every 3 months, dietitian visits every 3 months until meeting dietary recommendation or reaching 3 years limit, and daily tea drinking
  Interventions: Other: control:usual medical management; Behavioral: intervention 1:usual medical management+individual dieting consultation; Behavioral: intervention 2:usual medical management+individual dieting consultation+ daily tea drinking

INTERVENTIONS:
Other: control:usual medical management — with regular doctor visits every 3 months
Behavioral: intervention 1:usual medical management+individual dieting consultation — with regular doctor visits every 3 months and dietitian visits every 3 months
  Arms: usual medical management+individual dietary consultation; usual medical management+individual dietary consultation+ daily tea drinking
Behavioral: intervention 2:usual medical management+individual dieting consultation+ daily tea drinking — with regular doctor visits every 3 months and dietitian visits every 3 months and daily tea drinking
  Arms: usual medical management+individual dietary consultation+ daily tea drinking

SUMMARY:
Incidence of cardiometabolic disease (CMD) continues to rise, which consumes huge medical resources in Taiwan. The effectiveness of dietary therapy for CMD has not been locally evaluated in detail. CVD is an important risk factor for dementia. At the present time, there is no effective treatment available for dementia. Early prevention is extremely important. Our previous studies have shown that Taiwanese dementia protective diet is very similar to cardiovascular prevention and control diet, meaning that effective dietary therapy may not only control CVD but also prevent dementia development. Therefore, this study intends to document the effects of dietary intervention on cardiovascular disease risk factor control, the long-term outcomes on the occurrence of cardiovascular events, and the maintenance of cognitive function for patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

1. Have received percutaneous transluminal coronary artery surgery.
2. Stable drug control for more than one month

Exclusion Criteria:

1. Suffer from cancer and undergo chemotherapy or surgery within one year.
2. Those who have a major illness in hospital within one year.
3. Those with kidney disease stage 5 (inclusive) or above
4. Those whose life expectancy does not exceed half a year
5. Patients with diagnosed dementia
6. Those who do not want to be tracked

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-12-23 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline in diet quality at Year 1, 2, and 3. | Baseline, year 1, 2 and 3
  Diet quality is estimated according to the daily intake of nutrients and the distribution of the six food groups, with a qualified food frequency questionnaire.
  The six food groups include:
  1. Whole grains and starchy vegetables
  2. Protein foods: soybeans, fish, eggs, and meat
  3. Vegetables
  4. Fruits
  5. Dairy
  6. Oils, nuts & seeds
Change from baseline in concentrations of cardiovascular risk factors at Month 6, 12, 18, 24,30, and 36. | Baseline and Month 6, 12, 18, 24, 30, and 36.
  Cardiovascular risk factors include total cholesterol,triglyceride, low-density lipoprotein ,high-density lipoprotein, uric acid, glucose, HbA1C.
Events of cardiovascular diseases at Year 6. | Year 6.
  CVD or non-CVD death, stroke, acute myocardial infarction, hospitalization for acute coronary syndrome, hospitalization for coronary intervention surgery, hospitalization for various cardiovascular diseases, hospitalization for heart failure, hospitalization for other CVD diseases, new-onset heart arrhythmia, new-onset peripheral blood vessels block

SECONDARY OUTCOMES:
Change from baseline in the dosage of prescribed drugs at Month 6, 12, 18, 24,30, and 36. | Baseline and Month 6, 12, 18, 24, 30, and 36.
  Prescribed drugs for cardiovascular diseases.
Change from baseline in cardiovascular risk score | Baseline, year 1, 2 and 3.
  Taiwanese edition of Framingham Risk Score, a 10-year risk score derived as a percentage. Risk is considered low if the Framingham Risk Score is less than 10%, moderate if it is 10% to 19%, and high if it is 20% or higher.
Change from baseline in concentrations of inflammatory markers at Year 1, 2, and 3. | Baseline, year 1, 2 and 3.
  Inflammatory markers include IL-1β, IL-6, IL-8, IL-10，TNF- α, IFN-γ in blood.
Change from baseline in scores of Montreal Cognitive Assessment at Year 1, 2, and 3. | Baseline, year 1, 2 and 3.
  Scores on the Montreal Cognitive Assessment range from zero to 30. A score of 26 and higher is considered normal.
Change from baseline in scores of Number Cancellation test | Baseline, year 1, 2 and 3.
  A sub-scale of Alzheimer's Disease Assessment Scale. Cancellation score = number of targets hit in 45 seconds - (minus) number of errors - (minus) number of times reminded of the task.
Change from baseline in the number of digits at Year 1, 2 and 3. | Baseline, year 1, 2 and 3.
  A digit span task is used to measure working memory's number storage capacity. Subjects are read a sequence of numbers and asked to repeat the same sequence back to the examiner in order (forward span) or in reverse order (backward span). The score is the length of the longest correctly repeated sequence. The maximum number of digits in a sequence is 9 and the minimum number of digits in a sequence is 2. The higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Harn Pan, Ph.D, Principal Investigator — Institute of Biomedical Sciences, Academia Sinica
Locations (1):
- Taipei Veterans General Hospital, Taipei, Beitou District, Taiwan